CLINICAL TRIAL: NCT06837935
Title: Effect of Aluminum Foil Reflector on Phototherapy for Newborn Infants with Unconjugated Hyperbilirubinemia: a Randomized Controlled Trial
Brief Title: Aluminum Foil Reflector on Phototherapy for Newborn with Jaundice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202411028
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Newborn Jaundice
Keywords: Aluminum Foil Reflector; Phototherapy; Newborn; Hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aluminum Foil Reflector Group (Experimental): This group includes newborns who require phototherapy with an Aluminum Foil Reflector.
  Interventions: Device: Aluminum Foil Reflector
- Control group (No Intervention): This group includes newborns requiring phototherapy and not using an Aluminum Foil Reflector.

INTERVENTIONS:
Device: Aluminum Foil Reflector — The hyperbilirubinemia newborns will receive phototherapy with an Aluminum Foil Reflector around an incubator. The aluminum foil reflector, sewn inside a cloth that is 30 cm long and 3 mm thick, will be hung from the three sides of the phototherapy unit. The reflector will cover the whole incubator except for the foot part to allow infant observation during treatment. While receiving phototherapy, the lights will be continuously on, except during feeding, physical examination, and blood taking. All participants will dress only in nappies and eye masks during phototherapy treatment.
  Serum bilirubin will be taken every 24 hours until phototherapy can be stopped according to AAP guidelines.
  Arms: Aluminum Foil Reflector Group

SUMMARY:
Hyperbilirubinemia is defined as the presence of bilirubin in the serum of newborns at levels exceeding the normal range. It is the most common problem among healthy newborns, with an incidence of approximately 40% to 60% in full-term infants. The primary cause is the immature bilirubin metabolism in newborns, leading to the accumulation of excess bilirubin in the blood, which in turn results in a temporary yellowing of the skin and sclera, known as jaundice. Physiological jaundice in full-term newborns typically appears 24 to 72 hours after birth, peaking on days 4 to 5. Studies have shown that neonatal jaundice is a leading cause of readmission after discharge.

Phototherapy is the most effective and safest treatment for neonatal hyperbilirubinemia. It takes advantage of bilirubin's sensitivity to light, converting bilirubin into water-soluble conjugated bilirubin, which is then excreted through bile and urine, thereby reducing total bilirubin levels. The most effective light during phototherapy has a wavelength of 400 nm to 520 nm and an intensity of at least 30 microW/cm²/nm, with at least 80% of the infant's body surface area exposed.

This study aims to investigate whether using aluminum foil reflective covering around the phototherapy incubator can enhance the effectiveness of light treatment for jaundice in infants, thus potentially reducing the duration of phototherapy required.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns who are admitted to the neonatal ward for examination and treatment due to jaundice levels reaching the treatment threshold.
2. Term babies below 14 days of age (gestational age of 37 weeks or greater).
3. No evidence of hemolysis

Exclusion Criteria:

1. Infants with serum bilirubin levels close to the exchange transfusion limit
2. Hemolytic disease (Ex: G6PD)
3. Congenital anomalies
4. Elevated direct bilirubin
5. Infants with abnormal liver function or biliary structure
6. Infants who receive Cardiopulmonary Resuscitation after birth or suspected perinatal asphyxia

Ages: 1 Hour to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Decline in bilirubin | at 24 hours, 48 hours, 72 hours and the end of phototherapy
  The number of infants experiencing sufficient decline in bilirubin.
Phototherapy duration (hours) | From the date of beginning of phototherapy until the day of stop of phototherapy
  The total time of phototherapy, mean ± SD

SECONDARY OUTCOMES:
Bilirubinemia concentration | At 24 hours, 48 hours, 72 hours and the end of phototherapy
  Heel blood will be taken for serum bilirubin level assessment
Hospital stay (days) | From the hospitalization to the discharge of infants
  Number of days of hospital stay
Skin rash | From the beginning of phototherapy until the stop of phototherapy.
  Number of participants with redness, blisters, itchiness, and peeling.
Diarrhea | From the beginning of phototherapy until the stop of phototherapy.
  Number of participants having the signs of passing loose, watery stools three or more times a day

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Wai Tam, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuangho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No